CLINICAL TRIAL: NCT05177679
Title: Enhancing Children's Cognitive Function and Achievement Through Carotenoid Consumption
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Northeastern University (Other); University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21066
Record Dates: First submitted 2021-11-02; First posted 2022-01-04 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Cognitive Change; Achievement; Macular Pigmentation
Keywords: Lutein; Zeaxanthin; Carotenoids; Child; Spatial memory; Hippocampus; Academic success; Cognition

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Supplement (Experimental): The active supplementation group participants will be asked to consume a daily carotenoid supplement for 9 months.
  Interventions: Dietary Supplement: Active supplement
- Placebo Control (Placebo Comparator): The placebo control group participants will be asked to consume a placebo supplement for 9 months.
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Active supplement — Carotenoid supplement comprised of 10mg lutein and 2mg zeaxanthin.
  Arms: Active Supplement
Dietary Supplement: Placebo control — Placebo control supplement
  Arms: Placebo Control

SUMMARY:
The aim of this study is to test the casual relationship between carotenoid supplementation, cognitive function, and achievement over a school-year. The central hypothesis is that, relative to the waitlist placebo group, children receiving the carotenoid supplement will exhibit greater gains in cognitive function and achievement.

DETAILED DESCRIPTION:
This clinical trial will be a randomized placebo-controlled double-blind trial to examine the effects of carotenoid supplementation on cognitive control, hippocampal-dependent relational memory, and academic achievement among pre-adolescents over one school year (i.e. 9-months).

ELIGIBILITY:
Inclusion Criteria:

* Child assent and parent/guardian consent
* 8-10 years of age
* No lutein supplementation within 6-months prior to enrollment (exception of multivitamins containing less than 1 mg lutein/day)
* Absence of learning disability (parent-reported)
* Tanner scale score ≤ 2
* 20/20 or corrected vision

Exclusion Criteria:

* Non-assent of child or non-consent of guardian
* Above/below 8-10 years of age
* Lutein supplementation within 6-months prior to enrollment (including multivitamins containing more than 1 mg lutein/day)
* Identified learning disability (parent-reported)
* Tanner scale score > 2
* Not 20/20 or uncorrected vision

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 288 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Attentional Accuracy | 9 months (Baseline vs Follow-up)
  Changes in accuracy (%) between groups using a computerized flanker task.
Attentional Reaction Time | 9 months (Baseline vs Follow-up)
  Changes in reaction time (ms) between groups using a computerized flanker task.
Hippocampal-dependent Relational memory | 9 months (Baseline vs Follow-up)
  Spatial memory task accuracy
Composite Academic Achievement | 9 months (Baseline vs Follow-up)
  Kaufman Test of Academic and Educational Achievement II (KTEA III) composite or comprehensive academic achievement score. The scores are standard scores with a minimum score of 40 and a maximum score of 160 where a higher score indicates a better outcome.

SECONDARY OUTCOMES:
Macular Pigment Optical Density | 9 months (Baseline vs Follow-up)
  Changes in Macular Pigment Optical Density (log units) between groups using a macular densitometer.
Attentional Resource Allocation | 9 months (Baseline vs Follow-up)
  Changes in P3 event related potential amplitude (microvolts) between groups using a computerized flanker task.
Attentional Processing Speed | 9 months (Baseline vs Follow-up)
  Changes in P3 event related potential latency (ms) between groups using a computerized flanker task.
Math | 9 months (Baseline vs Follow-up)
  Assessed as Mass subtest standard scores on the KTEA III. The scores are standard scores with a minimum score of 40 and a maximum score of 160 where a higher score indicates a better outcome.
Reading | 9 months (Baseline vs Follow-up)
  Assessed as Reading subtest standard scores on the KTEA III. The scores are standard scores with a minimum score of 40 and a maximum score of 160 where a higher score indicates a better outcome.
Written Language | 9 months (Baseline vs Follow-up)
  Assessed as Written Language subtest standard scores on the KTEA III. The scores are standard scores with a minimum score of 40 and a maximum score of 160 where a higher score indicates a better outcome.
Reading Fluency | 9 months (Baseline vs Follow-up)
  Assessed as Reading Fluency subtest standard scores on the KTEA III. The scores are standard scores with a minimum score of 40 and a maximum score of 160 where a higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Naiman Khan, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (1):
- University of Illinois Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cannavale CN, Keye SA, Rosok L, Martell S, Holthaus TA, Reeser G, Raine LB, Mullen SP, Cohen NJ, Hillman CH, Hammond BR, Renzi-Hammond L, Khan NA. Enhancing children's cognitive function and achievement through carotenoid consumption: The Integrated Childhood Ocular Nutrition Study (iCONS) protocol. Contemp Clin Trials. 2022 Nov;122:106964. doi: 10.1016/j.cct.2022.106964. Epub 2022 Oct 15. PMID 36252934